CLINICAL TRIAL: NCT04900545
Title: Effect of Genetic Polymorphisms on Response to Beta Blocker Therapy in Egyptian Patients
Status: Completed | Type: Observational
Sponsor: Mohamed Saleh Fayed (Other)
Responsible Party: Sponsor-Investigator, Mohamed Saleh Fayed, Teaching assistant, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: PHCL135
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Acute Coronary Syndrome; Hypertension
MeSH Terms: conditions — Acute Coronary Syndrome; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be collected and stored in - 80°C environment for DNA extraction by DNA extraction kit according to manufacturer recommendation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- beta blocker navie patients with acute coronary syndrome

SUMMARY:
Beta-blockers represent a cornerstone for the treatment of coronary artery disease (CAD). Their protective effect is based on the negative inotropic and chronotropic features, which have been tested in a large number of randomized controlled trials, both in patients with myocardial infarction (MI) and in those with stable angina, demonstrating a reduction of adverse cardiovascular events, a relief of symptoms and a reduction of myocardial ischemia

However, considerable interpatient variability in response to β-blockers has been reported which indicates that a considerable proportion of β-blocker-treated patients do not achieve the warranted cardio protection with β- blockers. This highlights the importance of identifying biomarkers associated with variability in response to β-blockers to improve the current approach for β- blocker selection, which seems to be suboptimal.

This study aims to study the effect of polymorphism in adrenergic beta receptors on beta-blocker response in Egyptian patients.

ELIGIBILITY:
Inclusion Criteria:

1. Beta-blockers naïve patients
2. Patients been on beta-blocker therapy for at least 4 weeks.
3. Age (18-75) Years old.

Exclusion Criteria:

1. Non-Egyptians.
2. Kidney failure of any stage.
3. Liver failure of any stage.
4. Malignancy.
5. Pregnancy.
6. HR < 55 beats/min (in the absence of b-blocker therapy).
7. Presence of a cardiac pacemaker.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Beta-Blocker naive Egyptian patient with acute coronary syndrome.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Adrenergic receptors genes and blood pressure response to beta-blocker | Three months
  Investigate the association of the adrenergic receptor polymorphisms with reduction in blood pressure (expressed in units of millimeters of mercury "mmHg" ) in the Egyptian patients with acute coronary syndrome on beta blocker therapy.
Adrenergic receptors genes and heart rate response to beta-blocker | Three months
  Investigate the association of the adrenergic receptor polymorphisms with reduction in heart rate (expressed as beats per minute "BPM" ) in the Egyptian patients with acute coronary syndrome on beta blocker therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa A Sabry, PhD, Study Chair — Ains Shams university; Mohamed A Saleh, PhD, Study Director — Ain Shams University; Amal A EL-Kholy, PhD, Study Director — Ain Shams University; Mohamed S Fayed, Bsc, Principal Investigator — Ains Shams university
Locations (1):
- Ain Shams University Hospitals., Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided